CLINICAL TRIAL: NCT01016132
Title: Clinical Evaluation of a Silicone Hydrogel Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: P-019-C-055
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Results first posted 2011-01-12 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2011-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Device: lotrafilcon A contact lens — Investigational silicone hydrogel, single-vision, soft contact lens worn for four weeks at least as often as and on the same basis as participant's habitual lenses, as prescribed by participant's eye care practitioner -- ie., on a daily wear, flex wear, or extended wear basis.

SUMMARY:
The purpose of this study is to assess the performance of an investigational contact lens among contact lens wearers.

ELIGIBILITY:
Inclusion Criteria:

* Currently wearing lotrafilcon A lenses in both eyes for a minimum of 5 days per week, 8 hours per day, for 3 months.
* Removes contact lenses daily or sleeps overnight in contact lenses (up to 30 consecutive nights) as prescribed by regular eye care practitioner.
* Able to achieve distance visual acuity of at least 20/40 in each eye with study lenses.
* Other protocol inclusion/exclusion criteria may apply.

Exclusion Criteria:

* Eye injury or surgery within 12 months prior to enrollment.
* Currently enrolled in any clinical trial.
* History of corneal refractive surgery.
* Other protocol inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: In this single group study, all participants wore an investigational lotrafilcon A silicone hydrogel, single-vision, soft contact lens in both eyes for a period of four weeks. Participants wore the study lenses at least as often as they wore their habitual lenses, and as prescribed by their eye care practitioners -- ie., on a daily wear, flex wear, or extended wear basis.
Period: Overall Study
Arm/Group | All Participants
Started | 152
Completed | 151
Not Completed | 1
Not completed — Discomfort | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 152
Age Continuous [Mean (Standard Deviation); unit: years] | 33.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 55

OUTCOME MEASURES:

1. Primary Outcome: Overall Preference
Description: Overall preference when comparing study lenses to "habitual" lenses, as interpreted by the participant and reported on a questionnaire as a single, retrospective evaluation of four weeks' wear time. Overall preference was measured on a 5-point Likert scale as follows: Strongly Prefer Study Lenses; Somewhat Prefer Study Lenses; No Preference; Somewhat Prefer "Habitual" Lenses; Strongly Prefer "Habitual" Lenses.
Time Frame: 4 weeks of wear
Population: Analysis conducted per protocol, with exclusions due to reasons such as: major protocol deviations as determined by masked review; discontinuations; and/or missing responses.
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 145
Participants
  Strongly Prefer Study Lenses | 28
  Somewhat Prefer Study Lenses | 31
  NO Preference | 46
  Somewhat Prefer "Habitual" Lenses | 20
  Strongly Prefer "Habitual" Lenses | 20

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the trial: 49 days
Description: Individual exposure: four weeks
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/152
Other Adverse Events (participants affected / at risk) | 0/152

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.